CLINICAL TRIAL: NCT05223530
Title: Prenatal Programming of Childhood Obesity and Cardio Metabolic Disorders - Role of Maternal Obesity, Pregnancy Complications, and Maternal-fetal Metabolome
Brief Title: Prenatal Programming of Childhood Obesity and Cardio Metabolic Disorders
Status: Recruiting | Type: Observational
Sponsor: Helsinki University Central Hospital (Other)
Collaborators: University of Helsinki (Other); University of Oulu (Other); University of Edinburgh (Other)
Responsible Party: Principal Investigator, Saila Koivusalo, Principal Investigator, Helsinki University Central Hospital
Other Study IDs: HUS
Record Dates: First submitted 2022-01-18; First posted 2022-02-04 (Actual); Last update posted 2024-12-10 (Actual); Status verified 2024-12

CONDITIONS: Cardiometabolic Diseases; Obesity
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 7 Days
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Prevention of Pre-eclampsia and Intrauterine Growth Restriction (PREDO): The PREDO study is a cohort study that was started in 2005 in the Helsinki metropolitan area and Northern Karelia. In 2005-2009, it recruited a total of 4,777 women in the early pregnancy. Almost all subjects participated in stress monitoring during pregnancy. In addition, some mothers participated in either genetic, ultrasound, or drug research to develop methods for predicting and preventing pre-eclampsia and fetal growth retardation, and for identifying related factors.
  Some key objectives have been to determine whether the physical and mental well-being of the pregnant women could be relevant with hereditary factors for the course of pregnancy and the subsequent physical and mental development and health of the child.
  The previous follow-up phases have been performed 2 weeks and 6 months after the birth in 2006-2011 and at the age of approximately 2-6 and 7-12 years. More than 2,500 families participated in the most recent follow-up phase. Now it is 11-17 years of follow-up.
- Finnish Gestational Diabetes Prevention (RADIEL): The RADIEL study is a randomized multicenter study that was launched in 2008 in Helsinki, Espoo, Vantaa and Lappeenranta. Between 2008 and 2011, we recruited a total of 729 women for gestational diabetes prevention research. Subjects either planned to become pregnant or were in early pregnancy at the time of the study. Subjects were randomized to either receive diet and exercise intervention (active group) or to continue with normal counseling follow-up (control group). Study visits occurred every three months before pregnancy (if recruited before pregnancy), once in each trimester of pregnancy, and at 6 weeks, 6 months, and 12 months after delivery. The effectiveness of the intervention was measured with a variety of metrics.
  In 2013-2017, we invited mothers and children who participated in the RADIEL study to a 5-year follow-up of the project, and nearly 350 mother-child pairs participated. Now it is 11-17 years of follow-up.

SUMMARY:
This is a prospective 11-17 -years follow-up of two existing pregnancy cohort (PREDO) and prevention (RADIEL) studies. The main objective is to investigate the associations between maternal overweight, obesity, hypertensive disorders in pregnancy, gestational diabetes, and maternal-fetal metabolome, child's birth outcomes, and overweight and obesity and cardio metabolic health outcomes in childhood and adolescence. During this follow-up study, the mothers and their 11-17-year-old children are invited for a study visit and their cardio metabolic health is studied by many different methods.

DETAILED DESCRIPTION:
The study comprises two Finnish pregnancy cohort /prevention studies, in which mother-child pairs have already been followed from early pregnancy until the threshold of adolescence. During this project period the follow-up of PREDO and RADIEL mothers and children will be extended until 11-17 and 11-14 years of age, respectively. This adolescence follow-up will include detailed measurements of overweight/obesity, body composition, and cardiovascular and metabolic health as well as lifestyle factors.

Research methods:

1. Maternal cardiometabolic conditions during pregnancy (data available): is defined by maternal pre-pregnancy BMI extracted from the Medical Birth; gestational weight gain calculated from maternal weight at childbirth derived from antenatal cards; blood pressure and proteinuria from antenatal cards, and results of 2-h oral glucose tolerance test and diagnoses of gestational diabetes and hypertensive disorders (chronic hypertension, gestational hypertension, preeclampsia) extracted from medical records and verified by an expert jury comprising two medical doctors and a research nurse with expertise in obstetrics.
2. Maternal and fetal metabolome (data available): is quantified by using high-throughput proton nuclear magnetic resonance (NMR) metabolomics platform (Nightingale Health Ltd, Helsinki, Finland). In total 220 metabolites were quantified covering multiple metabolic pathways, including lipoprotein lipids and subclasses, apolipoproteins, fatty and amino acids, ketone bodies, glycolysis and gluconeogenesis-related metabolites, fluid balance and inflammation.
3. Child's overweight/obesity and cardiometabolic health in childhood (data available): Child's weight and height have been derived from the child health center registry with data available from birth to 7-11 years in PREDO and from birth to 5 years in RADIEL. The 24-h ambulatory blood pressure data are available in the PREDO study from the child follow-up at age 7-11 years, and in the RADIEL study from the 5-year follow-up visit.
4. Child's overweight/obesity and cardiometabolic health in adolescence (11-17yrs): (data entry and quality control 1/22-6/24) will include

   * Body weight, height, blood pressure, pulse
   * Tanner stage
   * Body fat percentage (bioimpedance, InBody)
   * Digital questionnaires: Background, and Assessment of the psychological development of the child: Child Behavior Checklist for Ages 6-18 (CBCL), Strengths and Difficulties Questionnaire (SDQ), and Sleep Disturbance Scale for Children (SDSC) substance abuse, Level of Puberty (Tanner scale), Food frequency questionnaire (FFQ)
   * ActiGraph (acceleration sensor), assessment of physical activity and sleep for 7 days
   * Blood samples for analyses of: glucose and insulin metabolism, vitamin D, Calcium, Phosphate, AFOS and PTH, blood samples for assessment of lipidomics and metabonomics, DNA-sample (blood and buccal) and samples for adipocytokines and inflammation marker assessment
   * Endothelial function and pulse wave velocity (PWV) will be assessed
   * An epigenome-wide association study (EWAS) will be performed in the offspring according to maternal obesity and GDM status.
   * Continuous glucose monitoring (CGM, Dexcom G6, Dexcom®, USA) will be assessed in a subpopulation of 150 children, aged 11-14 yrs: 50 overweight/obese and 50 normal weight children from high-risk pregnancies (RADIEL) and 50 normal weight controls form normal pregnancies (PREDO).
5. The following maternal data will be collected 11-17 years post partum (data entry and quality control 1/22-6/24):

   * Blood pressure, pulse, weight, height, BMI, waist and hip circumference
   * Body fat percentage (bioimpedance, InBody).
   * Laboratory tests: OGTT, insulin, glucose, HbA1c, ALAT, lipids, TSH, free T4, DNA sample (blood)
   * DNA sample from buccal mucosa
   * Spare blood for future analyses (metabonomics and lipidonomics studies, inflammatory markers incl, P-hCRP, P-IL-6, adiponectin, TNFa)
   * Digital questionnaires: background, diet (FFQ) and physical activity, psychological questionnaires: Center of Epidemiological Studies Depression Scale (CES-D), Beck Anxiety Inventory II (BDI-II), Pittsburgh Sleep Quality Index (PSQI), Cohen Perceived Stress Scale (PSS5), PANAS-10 (Positive and negative affect schedule), VAS Social Support (Visual Analogue Scale for Social Support), and STAI state (Spielberger State-Trait-Anxiety-Inventory-state version
   * food frequency questionnaire (FFQ)
   * ActiGraph (acceleration sensor), assessment of physical activity and sleep for 7 days
   * Endothelial function and pulse wave velocity (PWV)
6. National registries and patient records on the course of pregnancy, the growth and development of the child and related diseases or their risk factors

ELIGIBILITY:
Inclusion Criteria:

* all mothers participated originally in the PREDO or the RADIEL studies during pregnancy and with delivery during this index pregnancy

Exclusion Criteria:

-

Ages: 11 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Gender Based: Yes — Follow-up of pregnant women and their 11-17 year-old children
Study Population: The study population comprises two Finnish pregnancy cohort /prevention studies, in which mother-child pairs have already been followed from early pregnancy until the threshold of adolescence.
  Women for the PREDO study were enrolled at 12-14 gestational weeks and for the RADIEL study before conception or at 10-12 gestational weeks. They gave birth to a singleton live infant between 2006-2010 (PREDO) and 2008-2014 (RADIEL).
Sampling Method: Non-Probability Sample
Enrollment: 750 (Estimated)
Dates: Start 2022-02-25 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Body fat percentage | one measure at follow-up study visit:11-17 years after pregnancy
  Measured by Inbody 720 (bioimpedance)

SECONDARY OUTCOMES:
Blood pressure | 2-3 measurements at follow-up study visit: 11-17 years after pregnancy
  Both systolic and diastolic pressures are measured by Omron HBP-1320
Body mass index | one measure at follow-up study visit: 11-17 years after pregnancy
  weight (kg) / height (m)2
Pulse wave velocity | one measure at follow-up study visit: 11-17 years after pregnancy
  Measured by Complior Analyse, Alarm Medical
Time in target he percentage of time spent within the gestational diabetes glucose target range (<7,8 mmol/l) | 10 days measurements related to the 11-17 years follow-up study visit
  Dexcom G6 CGM (continuous glucose monitoring)
Body weight | one measurement at follow-up study visit: 11-17 years after pregnancy
  Measured with Seca Mod 878DR (scale)

CONTACTS AND LOCATIONS:
Locations (1):
- Saila Koivusalo, Helsinki, Finland